CLINICAL TRIAL: NCT02958475
Title: Mother's Milk Messaging: Evaluation of a Bilingual Application (APP) to Support Initiation and Exclusive Breastfeeding in New Mothers
Acronym: MMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: W.K. Kellogg Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-1740
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control (Experimental): Participants in control arm will receive normal standard messages about infant injury prevention.
  Interventions: Behavioral: Injury Prevention Messages
- Breastfeeding Messages plus Social Support (Active Comparator): Participant will receive between 5-7 text messages weekly through push notifications to their phone. The text messages are targeted at specific theoretical constructs such as outcome expectations/attitudes, barrier self-efficacy, reinforcing a message using peripheral (expert) opinion, eliciting a sense of social currency or providing a cue-to-action. In addition they will be able to download the MMM app, which will store text messages received. Additionally, participants in this arm will be able to link within the app to a private Facebook page. Participants can access this page through their app or directly via Facebook where they can view, comment, and share in response to posts. The MMM app has three main elements: text messages via push notification are stored and searchable on the app, access to a breastfeeding social support group on Facebook, and access to videos and written material to facilitate knowledge acquisition and skills building.
  Interventions: Behavioral: Social Support Group (Facebook); Behavioral: Breastfeeding messages
- Breastfeeding Messages only (Active Comparator): Participant will receive between 5-7 text messages weekly through push notifications to their phone. The text messages are targeted at specific theoretical constructs such as outcome expectations/attitudes, barrier self-efficacy, reinforcing a message using peripheral (expert) opinion, eliciting a sense of social currency or providing a cue-to-action.
  Interventions: Behavioral: Breastfeeding messages

INTERVENTIONS:
Behavioral: Social Support Group (Facebook) — The breastfeeding social support group on Facebook will be moderated to facilitate posting of shared experiences. Short videos, photographs, and written blurbs on related topics are posted on the Facebook page to reinforce the messaging and content of the texts.
  Arms: Breastfeeding Messages plus Social Support
Behavioral: Breastfeeding messages — The Mother's Milk Messaging app gives participants access to text messages via push notification on the app, as well as access to videos and written material to facilitate knowledge acquisition and skills building. The text messages are targeted at specific theoretical constructs such as outcome expectations/attitudes, barrier self-efficacy, reinforcing a message using peripheral (expert) opinion, eliciting a sense of social currency or providing a cue-to-action.
  Arms: Breastfeeding Messages only; Breastfeeding Messages plus Social Support
Behavioral: Injury Prevention Messages — The Mother's Milk Messaging app will provide participants in the control group with genetic injury prevention message.
  Arms: Attention Control

SUMMARY:
This study is being conducted to evaluate the breastfeeding support program utilizing bilingual English-Spanish tailored text messages and online support to support exclusive and continuous breastfeeding for new mothers--comparing texting alone, texting with an online support group to those with usual care. The cost involved in moderating the online groups and providing bidirectional consultation when needed will be evaluated and qualitative feedback from a subset of mothers in both intervention groups will be evaluated to determine what was effective, as well as suggestions for improvement of the messaging program.

DETAILED DESCRIPTION:
Women of child-bearing age are in the generation most likely to use texting to communicate, and most own a cellular phone, and that cell phones have been demonstrated to be efficacious in increasing Human Immunodeficiency Virus (HIV) medication compliance and smoking cessation, and in improving diabetes management, the investigators consider this may be a promising strategy to increase breastfeeding. The investigators developed theoretically-based text message content along with breast feeding informational and video content designed for delivery via closed private groups on social media based on formative work and then conducted a pilot study to text the effects of interactive messaging sent over a 12 week period (i.e. 6 weeks prior and after birth) that targeted barriers (e.g. insufficient milk, pain/sore nipples, breastfeeding in public, among others) on exclusivity and continuation of breastfeeding. The investigators innovative approach, called Mother's Milk Messaging (MMM) specifically targets low-income and minority mothers and has the potential to reach unprecedented numbers of mothers, to be standardized for later scalability, and to be cost-effective.

While Text4Baby texting application uses a similar approach, the text messages are not interactive and they do not address specific issues with breastfeeding. The device's social media content facilitates private, peer and expert support for breastfeeding in real time on a channel preferred by first time mothers.

Applying a theoretically-based framework, the investigators developed content stemming from Dr. Maya Bunik's previous published Breastfeeding Telephone Triage and Advice. Content was adapted for delivery via a mobile application (App) with attention to an Integrated Theory of mobile Health (mHealth) using best practices for app design for health promotion using social and mobile technology. The content was modified to facilitate engagement with content using technology, utilizing communication theories such as Gain and Loss Framing and Elaboration theory, and theories to support social networking and social support, along with behavioral health theories such as the Theory of Planned Behavior and Social Cognitive Theory.

The MMM app has three main elements: text messages via push notification are stored and searchable on the app, access to a breastfeeding social support group on Facebook, and access to videos and written material to facilitate knowledge acquisition and skills building. The text messages are targeted at specific theoretical constructs such as outcome expectations/attitudes, barrier self-efficacy, reinforcing a message using peripheral (expert) opinion, eliciting a sense of social currency or providing a cue-to-action. The breastfeeding social support group on Facebook will be moderated to facilitate posting of shared experiences. Short videos, photographs, and written blurbs on related topics are posted on the Facebook page to reinforce the messaging and content of the texts. After a successful pilot study of MMM the investigators are ready to test the benefits of supporting new mothers with breastfeeding using the investigators bilingual mobile phone application (app) and online support program.

ELIGIBILITY:
Inclusion Criteria:

* Women who are first time mothers
* Women ages 18-40
* Who can converse and write in English and/or Spanish
* Who reside in the U.S.
* Who are expecting a normal singleton birth
* Who are pregnant
* Have access to a computer connected to the Internet
* Have access to a mobile device that can receive text messages and access the Internet (smart phone)

Exclusion Criteria:

* Decisionally challenged

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Breastfeeding exclusivity | Baseline, 3 and 6 months
  Percent of exclusive feeds as a measured in the past 24 hrs (e.g. 80% breastmilk)

SECONDARY OUTCOMES:
Change in Breastfeeding Self-Efficacy Scale (BSES) | Baseline, 3 and 6 months
  Breastfeeding self-efficacy is very important variable in breastfeeding duration, as it predicts whether a mother chooses to breastfeed, how much effort she will put into it and how she will respond to breastfeeding related difficulties. Using the BSES Long form 33-item scale we will assess participants self-efficacy related to breastfeeding intention and duration.
Change in Iowa Infant Feeding Attitudes Scale (IIFAS) | Baseline, 3 and 6 months
  Assessing participants self-efficacy (confidence) toward infant feeding methods, The scale consists of 17 items, with items worded so that approximately half of the questions are favorable toward breast-feeding and the remaining questions favorable toward formula-feeding. These scores are then computed so that a high score reflects a preference for breast-feeding.
Change in Infant Feeding Intentions Scale (IFIS) | Baseline, 3 and 6 months
  To quantitatively assess strength of intentions to initiate breastfeeding and continue to provide breast milk as the sole source of milk throughout the first 6 months (as recommended by public health agencies).
Change in Infant Feeding Practices Survey II (IFPS-II) | Baseline, 3 and 6 months
  IFPS-II was a longitudinal study focusing on infant feeding practices throughout the first year of life and the diets of women in their 3rd trimester and at four months postpartum. Infant feeding behaviors include patterns of breastfeeding, formula feeding, solid food intake, and feeding other complementary foods and liquids. We will focus on assessing participants breastfeeding intention, attitudes and outcome expectancies.
Change in Social Support Questionnaire (SSQ6) | Baseline, 3 and 6 months
  The following questions ask about people in participant's life who provide them with help or support related to breastfeeding (family, friends, community).
Change in Perceived Breastfeeding Support Assessment Tool (PBSAT) | Baseline, 3 and 6 months
  A 29-item based two-dimensional tool that has acceptable psychometric properties, the PBSAT is context specific, comprehensive, and user-friendly, so it can be administered by health-care workers, employers, policy makers, and researchers to improve the quality of services of breast-feeding urban working mothers, and could ultimately improve child health.
The Bidirectional Acculturation Scale for Hispanic (BAS) | Baseline
  The Bidirectional Acculturation Scale for Hispanic (BAS) measures acculturation to both Hispanic and non-Hispanic culture. The BAS includes 24 items measuring acculturation to Hispanic culture and 12 items that measure Hispanic or non-Hispanic acculturation are divided as Language Use, Linguistic Proficiency and Electronic Media. Participants rate their agreement with statement about the frequency of their language use and their proficiency using a 4-point Likert type format.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Bunik, MD, MPH, Principal Investigator — Colorado School of Public Health; Jennifer Leiferman, PhD, Principal Investigator — Colorado School of Public Health; Sheana Bull, PhD MPH, Principal Investigator — Colorado School of Public Health
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bunik M, Dunn DM, Watkins L, Talmi A. Trifecta approach to breastfeeding: clinical care in the integrated mental health model. J Hum Lact. 2014 May;30(2):143-7. doi: 10.1177/0890334414523333. Epub 2014 Mar 4. PMID 24595703
- [Background] Holmes AV, McLeod AY, Bunik M. ABM Clinical Protocol #5: Peripartum breastfeeding management for the healthy mother and infant at term, revision 2013. Breastfeed Med. 2013 Dec;8(6):469-73. doi: 10.1089/bfm.2013.9979. PMID 24320091
- [Background] Jansson LM, Bunik M, Bogen DL. Lactation and the Marijuana-Using Mother. Breastfeed Med. 2015 Jul-Aug;10(6):342-3. doi: 10.1089/bfm.2015.0067. Epub 2015 Jun 29. No abstract available. PMID 26121013
- [Background] Neifert M, Bunik M. Overcoming clinical barriers to exclusive breastfeeding. Pediatr Clin North Am. 2013 Feb;60(1):115-45. doi: 10.1016/j.pcl.2012.10.001. PMID 23178062
- [Background] Neville MC, Anderson SM, McManaman JL, Badger TM, Bunik M, Contractor N, Crume T, Dabelea D, Donovan SM, Forman N, Frank DN, Friedman JE, German JB, Goldman A, Hadsell D, Hambidge M, Hinde K, Horseman ND, Hovey RC, Janoff E, Krebs NF, Lebrilla CB, Lemay DG, MacLean PS, Meier P, Morrow AL, Neu J, Nommsen-Rivers LA, Raiten DJ, Rijnkels M, Seewaldt V, Shur BD, VanHouten J, Williamson P. Lactation and neonatal nutrition: defining and refining the critical questions. J Mammary Gland Biol Neoplasia. 2012 Jun;17(2):167-88. doi: 10.1007/s10911-012-9261-5. Epub 2012 Jul 1. PMID 22752723
- [Background] Bunik M, Shobe P, O'Connor ME, Beaty B, Langendoerfer S, Crane L, Kempe A. Are 2 weeks of daily breastfeeding support insufficient to overcome the influences of formula? Acad Pediatr. 2010 Jan-Feb;10(1):21-8. doi: 10.1016/j.acap.2009.09.014. PMID 20129478
- [Background] Bunik M, Krebs NF, Beaty B, McClatchey M, Olds DL. Breastfeeding and WIC enrollment in the Nurse Family Partnership Program. Breastfeed Med. 2009 Sep;4(3):145-9. doi: 10.1089/bfm.2008.0140. PMID 19243262
- [Background] Bunik M, Clark L, Zimmer LM, Jimenez LM, O'Connor ME, Crane LA, Kempe A. Early infant feeding decisions in low-income Latinas. Breastfeed Med. 2006 Winter;1(4):225-35. doi: 10.1089/bfm.2006.1.225. PMID 17661603
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Fein SB, Labiner-Wolfe J, Scanlon KS, Grummer-Strawn LM. Selected complementary feeding practices and their association with maternal education. Pediatrics. 2008 Oct;122 Suppl 2:S91-7. doi: 10.1542/peds.2008-1315l. PMID 18829837
- [Background] Noel-Weiss J, Boersma S, Kujawa-Myles S. Questioning current definitions for breastfeeding research. Int Breastfeed J. 2012 Aug 13;7(1):9. doi: 10.1186/1746-4358-7-9. PMID 22889093
- [Background] Nommsen-Rivers LA, Dewey KG. Development and validation of the infant feeding intentions scale. Matern Child Health J. 2009 May;13(3):334-42. doi: 10.1007/s10995-008-0356-y. Epub 2008 May 13. PMID 18473131